CLINICAL TRIAL: NCT01731015
Title: A Pilot Study for Evaluation of Regional Lung Function in Normal Subjects and Subjects With Airway and Lung Disorders Using 1H Magnetic Resonance Imaging With Oxygen as a Contrast Agent
Brief Title: Imaging Lung Function Using Oxygen Enhanced MRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hal C Charles (Other)
Responsible Party: Sponsor-Investigator, Hal C Charles, Associate Professor Department of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00024828; DIAL1001002 (Other: Duke University Medical Center)
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2012-11

CONDITIONS: COPD; Asthma; Cystic Fibrosis; Emphysema; Small Airways Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Cystic Fibrosis; Emphysema | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Subject (Experimental): Each subject will receive oxygen as a contrast agent to visualize the airway and alveolar spaces in their lungs using magnetic resonance imaging of inert gas/oxygen mixtures. The subjects will receive the gas by breathing room air interleaved with oxygen using a standard Douglas Bag system. No additional drug products, investigational or otherwise will be provided in this study.
  Interventions: Drug: Medical Grade Oxygen
- Subjects with Lung/or Airway Disease (Experimental): Each subject will receive oxygen as a contrast agent to visualize the airway and alveolar spaces in their lungs using magnetic resonance imaging of inert gas/oxygen mixtures. The subjects will receive the gas by breathing room air interleaved with oxygen using a standard Douglas Bag system. No additional drug products, investigational or otherwise will be provided in this study.
  Interventions: Drug: Medical Grade Oxygen

INTERVENTIONS:
Drug: Medical Grade Oxygen — At the study visits, MRI 'studies' will be performed using the same MR scanner (a 3.0-Tesla (T) TRIO MRI system (Siemens Medical Systems)). Lung morphology and function will be acquired using conventional 1H MRI followed by 1H MRI with oxygen as a gaseous contrast agent. For both series the subject will lie down in a supine position on the magnet bed with a standard 1H Torso coil for imaging. Subjects are scanned on room air and then the subjects are switched from room air to 100% oxygen and exhaled O2/CO2 are monitored (Oxigraf Capnograph) until steady state is achieved (in our experience ~ 1-2 minutes). The 100% oxygen MRI imaging is commenced (the average exposure time is usually 5-6 minutes with a maximum exposure of 15 minutes) after which the subjects are switched to room air. After steady state is achieved a second room air scan is completed.
  Other Names: oxygen

SUMMARY:
The goal of this study is to perform a pilot study to evaluate the utilization of oxygen as an inhaled contrast agent to image the airway spaces in normal and diseased human lungs to allow an effect size estimate to power future studies.

DETAILED DESCRIPTION:
This is an open label study expanding on work by other groups in animals, ex-vivo human lungs and human subjects. Both 2-dimensional and 3-dimensional images will be obtained using 1H MRI comparing images obtained while breathing oxygen to those obtained breathing room air.

Objectives

* To determine if 1H magnetic resonance images of the human lung and airways can be obtained in both single breath-hold and gated breathing imaging studies with adequate signal level and image contrast to extract regional lung functional information with oxygen as a contrast agent.
* To determine the short term reproducibility of the lung functional imaging in a subset of subjects (5 control subjects and 5 subjects with lung disease) with repeat MRI studies (Visit 2) at a time point ≥ 1 week to ≤ 4 weeks from Visit 1

ELIGIBILITY:
Inclusion Criteria for Lung and/or Airway Disease

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

  1. Subjects must be ≥ 18 years of age;
  2. Evidence of lung disease or injury by medical history, physical exam, and/or clinical laboratories;

     * COPD
     * Asthma
     * Pre/Post Lung Transplant
     * Cystic Fibrosis
     * Emphysema/Other Small Airways Diseases
     * Lung Transplant
  3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
  4. Subjects who are willing and able to comply with scheduled visits and other trial procedures.

Exclusion Criteria for Subjects with Lung and/or Airway Disease:

Subjects presenting with any of the following will not be included in the trial:

1. Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications (e.g. metal in the eye, claustrophobia);
2. Unable to receive 100% oxygen by breathing because of potential hypercapnia ( SpO2 <90% or FEV1 < 1 L);
3. Participation in a clinical trial with a study drug that may impact lung function in the past 14 days; or
4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial. This determination is made by the referring physician based on standard clinical practice.
5. Female; women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MR scan, prior to the MRI scan.

Inclusion Criteria for Normal Subjects Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Subjects must be ≥ 18 years of age;
2. Non-smokers, ex-smokers with normal pulmonary function test by spirometry;
3. No Evidence of prior lung disease or lung injury by medical history, physical exam, and/or clinical laboratories;
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
5. Subjects who are willing and able to comply with scheduled visits and other trial procedures.

Exclusion Criteria for Normal Subjects

Subjects presenting with any of the following will not be included in the trial:

1. Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications (e.g. metal in the eye, claustrophobia);
2. Unable to receive 100% oxygen by breathing because of potential hypercapnia (SpO2 <90% or FEV1 < 1 L) (Note, we consider this highly unlikely in a 'normal' subject);
3. Participation in a clinical trial with a study drug that may impact lung function in the past 14 days; or
4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
5. Female; women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MR scan, prior to the MRI scan.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Image Quality | one exposure
  Assessment of image quality of oxygen enhanced MR images: Signal to Noise Ratio, Dynamic Range of Ratio/Difference Images

CONTACTS AND LOCATIONS:
Overall Officials: Cecil Charles, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States